CLINICAL TRIAL: NCT06197334
Title: Gastro-intestinal Biopotential Recorder by Means of Surface ELEctrodes
Acronym: GRELE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CARON Bénédicte, MD, PhD, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A01618-37
Record Dates: First submitted 2023-12-19; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease; Functional Gastrointestinal Disorders; Healthy
Keywords: Medical device; Electrophysiology
MeSH Terms: conditions — Crohn Disease; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteers (Experimental)
  Interventions: Device: Gastro-intestinal biopotentials recording
- Crohn's disease patients with fibrosis (Experimental)
  Interventions: Device: Gastro-intestinal biopotentials recording
- Crohn's disease patients without fibrosis (Experimental)
  Interventions: Device: Gastro-intestinal biopotentials recording
- Functional gastrointestinal disorders patients (Experimental)
  Interventions: Device: Gastro-intestinal biopotentials recording

INTERVENTIONS:
Device: Gastro-intestinal biopotentials recording — Participants will undertake two recordings made with the device. The first one will last 1 hour and 30 minutes and will occurs while the participants are fasting. Then, they will eat a standardized meal. Finally, the second recording will take place after the meal ingestion and will last 1 hour and 30 minutes while the participants are in postprandial state.

SUMMARY:
The goal of this clinical trial is to compare the gastro-intestinal biopotentials recorded with a homemade device using surface electrodes placed on the abdomen in healthy volunteers, Crohn's disease patients without fibrosis, Crohn's disease patients with fibrosis and in functional gastrointestinal disorders (FGID) patients.

The main question it aims to answer is:

• Is there any differences in the gastro-intestinal biopotentials between the different populations under study?

It aims to answer two secondary questions:

* Are the gastro-intestinal biopotentials comparable to the Harvey-Bradshaw Index, MRI and biological data for patients with Crohn's disease?
* Are the gastro-intestinal biopotentials comparable to Rome IV criteria for functional gastrointestinal disorders patients?

Participants will undertake two recordings made with the device. The first one will last 1 hour and 30 minutes and will occurs while the participants are fasting. Then, the participants will eat a standardized meal. Finally, the second recording will take place after the meal ingestion and will last 1 hour and 30 minutes while the participants are in postprandial state.

DETAILED DESCRIPTION:
Diseases and disorders of the digestive tract affect a large proportion of the world's population. These disorders or diseases degrade patients' quality of life and are costly for healthcare systems. Today, it is difficult to categorize, monitor and/or prognosticate their evolution due to their unknown etiologies, the long duration of the digestion processes and unsuitable (invasive, complex or costly) examinations.

However, electrophysiology holds great promise for the study of these diseases. Indeed, the organs of the digestive tract are made up of longitudinal and circular muscles which contract rhythmically and synchronously to advance the food bolus during digestion, or to cleanse the digestive tract once digestion is complete.

No study has yet demonstrated the feasibility and value of measuring these bio-potentials for Functional Gastro Intestinal Disorders and Inflammatory Bowel Diseases.

That's why a homemade gastro-intestinal biopotentials recorder was developped. The recorder uses surface electrodes placed on the abdomen to record this biopotentials. The investigators hypothesize that surface gastro-intestinal biopotentials differ between a population of healthy volunteers, Crohn's disease patients and FGID patients.

ELIGIBILITY:
Inclusion Criteria for all participants:

* Person age > 18 years
* Person has been fasting for at least 12 hours
* Person who has received full information on the organization of the research and has not objected to the use of this data.
* Person affiliated to or beneficiary of a social security plan
* Person informed about study organization and having signed the informed consent

Inclusion Criteria for healthy volunteers :

* Person has no history of chronic gastro-intestinal disease
* Person has no acute of gastro-intestinal disease

Inclusion Criteria for Crohn's disease patients without fibrosis :

* Person is already diagnosed with Crohn's disease
* Person has underwent during the last 6 months :
* An MRI showing no fibrosis
* A blood test for C-reactive protein and fecal calprotectine
* A questionnaire to asses the Harvey-Bradshaw Index

Inclusion Criteria for Crohn's disease patients with fibrosis :

* Person is already diagnosed with Crohn's disease
* Person has underwent during the last 6 months :
* An MRI showing fibrosis
* A blood test for C-reactive protein and fecal calprotectine
* A questionnaire to asses the Harvey-Bradshaw Index

Inclusion Criteria for functional gastrointestinal disorders patients :

* Person is already diagnosed with functional gastrointestinal disorders
* Person has underwent an evaluation of the Rome IV criteria

Exclusion Criteria for all participants:

* Person having a pacemaker
* Person suffering from a sensory disorder making insensitive to pain on the skin
* Person suffering from a mental or motor disorders creating uncontroled movements
* Person being allergic to one or more component of the device
* Person being allergic to : soy, dairy food, peanuts, wheat, nuts
* Person having an history of gastro-intestinal surgery
* Person suffering from injury or erythema on the abdominal skin
* Person having a contagious potential (bacterial, fungal or viral)
* Person being in menstruation period
* Person suffering from urinary incontinence
* Minor (not emancipated)
* Person of legal age (subject to a legal protection measure)
* Adult unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Gastro-intestinal biopotentials pattern as recorded by the homemade recorder | 12 months
  Gastro-intestinal biopotentials pattern in patients versus healthy volunteers

SECONDARY OUTCOMES:
Correlation score between gastro-intestinal biopotentials pattern as recorded by the homemade recorder vs Harvey-Bradshaw Index assessed with a questionnaire | 12 months
  Correlation score in Crohn's disease patients with and without fibrosis for the gastro-intestinal biopotentials pattern vs the Harvey-Bradshaw Index
Correlation score between gastro-intestinal biopotentials pattern as recorded by the homemade recorder vs the Nancy score assessed by a clinician rating MRI images | 12 months
  Correlation score in Crohn's disease patients with and without fibrosis for the gastro-intestinal biopotentials pattern vs the Nancy score (MRI score)
Correlation score between gastro-intestinal biopotentials pattern as recorded by the homemade recorder vs blood fecal calprotectin levels (µg/g) | 12 months
  Correlation score in Crohn's disease patients with and without fibrosis for the gastro-intestinal biopotentials pattern vs blood fecal calprotectin levels
Correlation score between gastro-intestinal biopotentials pattern as recorded by the homemade recorder vs C-reactive protein levels (µg/L) | 12 months
  Correlation score in Crohn's disease patients with and without fibrosis for the gastro-intestinal biopotentials pattern vs C-reactive protein levels
Correlation score between gastro-intestinal biopotentials pattern as recorded by the homemade recorder vs Rome IV criteria | 12 months
  Correlation score in functional gastrointestinal disorders patients for the gastro-intestinal biopotentials pattern vs the Rome IV criteria

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy - Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alighaleh S, Cheng L, Angeli-Gordon TR, Aghababaie Z, O'Grady G, Paskaranandavadivel N. Design and Validation of a Surface-Contact Electrode for Gastric Pacing and Concurrent Slow-Wave Mapping. IEEE Trans Biomed Eng. 2021 Aug;68(8):2574-2581. doi: 10.1109/TBME.2021.3063685. Epub 2021 Jul 16. PMID 33656985
- [Background] Axelrod L, Axelrod S, Navalgund A, Triadafilopoulos G. Pilot Validation of a New Wireless Patch System as an Ambulatory, Noninvasive Tool That Measures Gut Myoelectrical Signals: Physiologic and Disease Correlations. Dig Dis Sci. 2021 Oct;66(10):3505-3515. doi: 10.1007/s10620-020-06663-y. Epub 2020 Oct 15. PMID 33063188
- [Background] Bassotti G, Antonelli E, Villanacci V, Salemme M, Coppola M, Annese V. Gastrointestinal motility disorders in inflammatory bowel diseases. World J Gastroenterol. 2014 Jan 7;20(1):37-44. doi: 10.3748/wjg.v20.i1.37. PMID 24415856
- [Background] Calder S, Cheng LK, Andrews CN, Paskaranandavadivel N, Waite S, Alighaleh S, Erickson JC, Gharibans A, O'Grady G, Du P. Validation of noninvasive body-surface gastric mapping for detecting gastric slow-wave spatiotemporal features by simultaneous serosal mapping in porcine. Am J Physiol Gastrointest Liver Physiol. 2022 Oct 1;323(4):G295-G305. doi: 10.1152/ajpgi.00049.2022. Epub 2022 Aug 2. PMID 35916432
- [Background] Erickson JC, Bruce LE, Taylor A, Richman J, Higgins C, Wells CI, O'Grady G. Electrocolonography: Non-Invasive Detection of Colonic Cyclic Motor Activity From Multielectrode Body Surface Recordings. IEEE Trans Biomed Eng. 2020 Jun;67(6):1628-1637. doi: 10.1109/TBME.2019.2941851. Epub 2019 Sep 16. PMID 31535980
- [Background] Gharibans AA, Hayes TCL, Carson DA, Calder S, Varghese C, Du P, Yarmut Y, Waite S, Keane C, Woodhead JST, Andrews CN, O'Grady G. A novel scalable electrode array and system for non-invasively assessing gastric function using flexible electronics. Neurogastroenterol Motil. 2023 Feb;35(2):e14418. doi: 10.1111/nmo.14418. Epub 2022 Jun 14. PMID 35699340
- [Background] Huizinga JD, Lammers WJ. Gut peristalsis is governed by a multitude of cooperating mechanisms. Am J Physiol Gastrointest Liver Physiol. 2009 Jan;296(1):G1-8. doi: 10.1152/ajpgi.90380.2008. Epub 2008 Nov 6. PMID 18988693
- [Background] Khan, M.U., Aziz, S., Sohail, M., Shahid, A.A., Samer, S., 2019. Automated Detection and Classification of Gastrointestinal Diseases using surface-EMG Signals, in: 2019 22nd International Multitopic Conference (INMIC). IEEE, pp. 1-8. https://doi.org/10.1109/INMIC48123.2019.9022741
- [Background] Navalgund, A., Axelrod, S., Triadafilopoulos, G., 2015. Feasibility of measuring the contractile electrical complex over 72 hours in a healthy human subject using a wearable, wireless electrode patch.
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Peery AF, Crockett SD, Murphy CC, Lund JL, Dellon ES, Williams JL, Jensen ET, Shaheen NJ, Barritt AS, Lieber SR, Kochar B, Barnes EL, Fan YC, Pate V, Galanko J, Baron TH, Sandler RS. Burden and Cost of Gastrointestinal, Liver, and Pancreatic Diseases in the United States: Update 2018. Gastroenterology. 2019 Jan;156(1):254-272.e11. doi: 10.1053/j.gastro.2018.08.063. Epub 2018 Oct 10. PMID 30315778
- [Background] Riezzo G, Russo F, Indrio F. Electrogastrography in adults and children: the strength, pitfalls, and clinical significance of the cutaneous recording of the gastric electrical activity. Biomed Res Int. 2013;2013:282757. doi: 10.1155/2013/282757. Epub 2013 May 25. PMID 23762836
- [Background] Sperber AD, Bangdiwala SI, Drossman DA, Ghoshal UC, Simren M, Tack J, Whitehead WE, Dumitrascu DL, Fang X, Fukudo S, Kellow J, Okeke E, Quigley EMM, Schmulson M, Whorwell P, Archampong T, Adibi P, Andresen V, Benninga MA, Bonaz B, Bor S, Fernandez LB, Choi SC, Corazziari ES, Francisconi C, Hani A, Lazebnik L, Lee YY, Mulak A, Rahman MM, Santos J, Setshedi M, Syam AF, Vanner S, Wong RK, Lopez-Colombo A, Costa V, Dickman R, Kanazawa M, Keshteli AH, Khatun R, Maleki I, Poitras P, Pratap N, Stefanyuk O, Thomson S, Zeevenhooven J, Palsson OS. Worldwide Prevalence and Burden of Functional Gastrointestinal Disorders, Results of Rome Foundation Global Study. Gastroenterology. 2021 Jan;160(1):99-114.e3. doi: 10.1053/j.gastro.2020.04.014. Epub 2020 Apr 12. PMID 32294476
- [Background] Gharibans AA, Coleman TP, Mousa H, Kunkel DC. Spatial Patterns From High-Resolution Electrogastrography Correlate With Severity of Symptoms in Patients With Functional Dyspepsia and Gastroparesis. Clin Gastroenterol Hepatol. 2019 Dec;17(13):2668-2677. doi: 10.1016/j.cgh.2019.04.039. Epub 2019 Apr 19. PMID 31009794